CLINICAL TRIAL: NCT01412736
Title: A Phase IIa , Double-blind, Placebo-controlled Dose-ranging Study to Evaluate the Efficacy and Safety of KHK4563 in Adults With Uncontrolled, Suspected Eosinophilic Asthma
Brief Title: A Phase IIa Study of KHK4563
Acronym: 4563-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4563-003
Record Dates: First submitted 2011-08-07; First posted 2011-08-09 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Uncontrolled and Suspected Eosinophilic Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2mg (Experimental): sterile lyophilized formulation, 2mg
  Interventions: Drug: KHK4563
- 20mg (Experimental): sterile lyophilized formulation, 20mg
  Interventions: Drug: KHK4563
- 100mg (Experimental): sterile lyophilized formulation, 100mg
  Interventions: Drug: KHK4563
- Placebo (Placebo Comparator): two SC administration on day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK4563 — every 4 weeks for the first 3 doses on Weeks 0 (Day 1), 4, and 8 and then every 8 weeks thereafter for the last 4 doses on Weeks 16, 24, 32, and 40.
  Arms: 2mg
Drug: KHK4563 — every 4 weeks for the first 3 doses on Weeks 0 (Day 1), 4, and 8 and then every 8 weeks thereafter for the last 4 doses on Weeks 16, 24, 32, and 40.
  Arms: 20mg
Drug: KHK4563 — every 4 weeks for the first 3 doses on Weeks 0 (Day 1), 4, and 8 and then every 8 weeks thereafter for the last 4 doses on Weeks 16, 24, 32, and 40.
  Arms: 100mg
Drug: Placebo — every 4 weeks for the first 3 doses on Weeks 0 (Day 1), 4, and 8 and then every 8 weeks thereafter for the last 4 doses on Weeks 16, 24, 32, and 40.
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled dose-ranging study of KHK4563 to evaluate the effect of multiple-dose subcutaneous administration of KHK4563 on the annual asthma exacerbation rate in adult subjects with uncontrolled, suspected eosinophilic asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 through 75 years at the time of Week -3 visit.
2. Written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
3. Physician prescribed daily use of medium-dose or high-dose ICS plus LABA or any combination of sequential dosing of either medium-dose or high-dose ICS/LABA for at least 12 months prior to Week -3 visit. Dose must be stable for at least 30 days prior to Week -3 visit.
4. At least 2, but not more than 6, documented asthma exacerbations in the 12 months prior to Week -3 visit that required use of a systemic corticosteroid burst.

Exclusion Criteria

1. Any condition (eg, any eosinophilic lower respiratory disease other than asthma, Churg-Strauss syndrome, hypereosinophilic syndrome, eosinophilic bronchitis, eosinophilic pneumonia, chronic obstructive pulmonary disease (COPD), bronchiectasis or cystic fibrosis (CF)) that, in the opinion of the investigator or Medical Expert, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
2. Any clinically relevant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis during screening period, which in the opinion of the investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to participate in the study.
3. Acute upper or lower respiratory infections requiring antibiotics or antiviral medications within 30 days prior to Week -3 visit or during the screening period.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
evaluation of the effect of multiple-dose subcutaneous(SC) administration of benralizumab on the annual asthma exacerbation rate in adult subjects with uncontrolled, suspected eosinophilic asthma. | Immediately following the first administration of study drug through Study Week 52.
  annual asthma exacerbation rate

SECONDARY OUTCOMES:
Pulmonary function as assessed by Forced Expiratory Volume in 1 Second (FEV1) and Peak Expiratory flow (PEF) | From first administration of study drug through Study Week 52.
  Pre-dose/pre-bronchodilator Forced Expiratory Volume in 1 Second ( FEV1 ) at the study centre, morning and evening peak expiratory flow (PEF)
Asthma control as assessed by ASTHMA CONTROL QUESTIONNAIRE6(ACQ6) | From first administration of study drug through Study Week 52.
  ASTHMA CONTROL QUESTIONNAIRE6(ACQ6)
Number of participants with Adverse Events as a Measure of Safety and Tolerability | From first administration of study drug through Study Week 68.
  Adverse Events/Serious Adverse Events (AE/SAE) - Laboratory variables - ECG (Electrocardiogram) - Physical Examination
Time Profiles of Serum Concentration | From first administration of study drug through Study Week 68
  Serum benralizumab concentration
Immunogenicity by serum incidence rate of positive anti-drug antibody | From first administration of study drug through Study Week 68
  Anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Locations (29):
- Japan (24):
  - Nagoya, Aichi-ken
  - Toyota-shi, Aichi-ken
  - Kamogawa-shi, Chiba
  - Fukuoka, Fukuoka
  - Ogaki-shi, Gifu
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Himeji-shi, Hyōgo
  - Kobe, Hyōgo
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Nagasaki, Nagasaki
  - Kishiwada-shi, Osaka
  - Koshigaya-shi, Saitama
  - Shizuoka, Shizuoka
  - Itabashi-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Mizunami-shi
  - Osakasayama-shi
  - Oura-gun
  - Seto-shi
- South Korea (5):
  - Chungcheongbuk-do
  - Gwangju
  - Gyenggi-do
  - Seoul
  - Suwon